CLINICAL TRIAL: NCT00000287
Title: Relapse Patterns in Female Cocaine Users
Brief Title: Relapse Patterns in Female Cocaine Users - 4
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Other Study IDs: NIDA-09259-4; P50-09259-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders

SUMMARY:
The purpose of this study is to pilot a relapse questionnaire and examine relapse patterns in female cocaine users.

DETAILED DESCRIPTION:
The objectives of this study were to determine the most important antecedent factors in relapse episodes and difference in the use of coping skills between relapses and "close calls"

ELIGIBILITY:
Inclusion Criteria:

Female, cocaine abuse or dependency by SCIS, at least 7 days of current abstinence, cocaine use of 8 out of 30 days prior to current abstinence, ages 18-60.

Exclusion Criteria:

Inability to participate in a 90 day longitudinal study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1995-02; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Presented at CPDD 1995 and ASAM 1997. Presented at CPDD 1995 and ASAM 1997.